CLINICAL TRIAL: NCT00002514
Title: Phase III Randomized Trial of Autologous and Allogeneic Stem Cell Transplantation Versus Intensive Conventional Chemotherapy in Acute Lymphoblastic Leukemia in First Remission
Brief Title: Stem Cell Transplantation Compared With Standard Chemotherapy in Treating Patients With Acute Lymphoblastic Leukemia in First Remission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000078099; E2993; MRC-LEUK-UKALL-XII; EST-4491; NCT00222586 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Leukemia
Keywords: adult acute lymphoblastic leukemia in remission
MeSH Terms: conditions — Leukemia | interventions — sargramostim; Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Etoposide; Imatinib Mesylate; Leucovorin; Mercaptopurine; Methotrexate; Prednisone; Thioguanine; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transplant (Experimental): Allogeneic (if donor) or Autologous (if no donor) bone marrow transplant
  Interventions: Biological: sargramostim; Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: etoposide; Drug: imatinib mesylate; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: vincristine sulfate; Procedure: allogeneic bone marrow transplantation; Procedure: autologous bone marrow transplantation; Procedure: peripheral blood stem cell transplantation
- Conventional Consolidation/Maintenance (Active Comparator): Consolidation/Maintenance Therapy
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: etoposide; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Biological: sargramostim
  Arms: Transplant
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
  Arms: Conventional Consolidation/Maintenance
Drug: etoposide
Drug: imatinib mesylate
  Arms: Transplant
Drug: leucovorin calcium
Drug: mercaptopurine
Drug: methotrexate
Drug: prednisone
Drug: thioguanine
  Arms: Conventional Consolidation/Maintenance
Drug: vincristine sulfate
Procedure: allogeneic bone marrow transplantation
  Arms: Transplant
Procedure: autologous bone marrow transplantation
  Arms: Transplant
Procedure: peripheral blood stem cell transplantation
  Arms: Transplant
Radiation: radiation therapy
  Arms: Conventional Consolidation/Maintenance

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with allogeneic or autologous stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. It is not yet known whether stem cell transplantation is more effective than standard chemotherapy in treating acute lymphoblastic leukemia.

PURPOSE: This randomized phase III trial is studying how well stem cell transplantation works compared to standard combination chemotherapy in treating patients with acute lymphoblastic leukemia in first remission.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the duration of complete remission (CR) and survival in patients with acute lymphoblastic leukemia in first remission treated with allogeneic or autologous stem cell transplantation (SCT) vs conventional consolidation and maintenance chemotherapy.
* Compare the overall treatment outcomes in patients treated with these regimens.
* Determine the effect of imatinib mesylate given after induction therapy in Philadelphia (Ph) chromosome-positive patients in CR.
* Determine the benefit of allogeneic or autologous SCT after imatinib mesylate in Ph chromosome-positive patients.
* Determine the benefit of additional imatinib mesylate administered after allogeneic or autologous SCT in Ph chromosome-positive patients.
* Determine the minimal residual disease in Ph chromosome-positive patients before and after treatment with imatinib mesylate.
* Determine the clinical resistance to imatinib mesylate caused by BCR-ABL gene amplification or mutation in Ph chromosome-positive patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (50 and under vs over 50), time to achieve complete remission (CR) (4 weeks or less vs more than 4 weeks), and Philadelphia (Ph) chromosome status (positive vs negative).

* First induction therapy: Patients receive daunorubicin (DNR) IV over 15-30 minutes and vincristine (VCR) IV over 3-5 minutes on days 1, 8, 15, and 22; oral prednisone (PRED) once daily on days 1-28; and asparaginase (ASP) IV over 30 minutes or intramuscularly on days 17-28. Patients with CNS leukemia at presentation also receive methotrexate (MTX) intrathecally (IT) via an Ommaya reservoir weekly until the CSF is clear. Patients without CNS leukemia at presentation receive MTX IT on day 23 only.
* Second induction therapy: Beginning immediately after first induction therapy, patients receive cyclophosphamide (CTX) IV over 30 minutes on days 1, 15, and 29; cytarabine (ARA-C) IV over 30 minutes on days 1-4, 8-11, 15-18, and 22-25; and oral mercaptopurine (MP) once daily on days 1-28. Patients with CNS leukemia at presentation also undergo concurrent craniospinal irradiation. Patients without CNS leukemia at presentation receive MTX IT on days 1, 8, 15, and 22. Patients with Ph chromosome-positive status receive oral imatinib mesylate once daily for at least 28 days (days 1-28).

Patients with Ph chromosome-positive status and CR after second induction therapy proceed to group I for autologous or allogeneic stem cell transplantation (SCT). Patients with Ph chromosome-negative status and CR after second induction therapy proceed to group II.

* Group I (Ph chromosome-positive patients):

  * Autologous SCT: Patients receive high-dose consolidation/mobilization chemotherapy comprising ARA-C IV over 3 hours on days 1-3 and mitoxantrone IV immediately after ARA-C administration on days 1 and 2. Patients also receive filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 5 and continuing until blood counts recover.

Patients then undergo peripheral blood stem cell collection or bone marrow harvesting.

Patients receive preparative therapy comprising total body irradiation twice daily (5-10 hours apart) on days -6 to -4 and high-dose etoposide (VP-16) IV over 4 hours on day -3. Male patients also undergo radiotherapy boost to the testes on day -6.

Patients undergo autologous SCT on day 0 and receive sargramostim (GM-CSF) SC once daily beginning 6 hours after the completion of SCT and continuing until blood counts recover.

* Allogeneic SCT: Patients receive the preparative regimen as in autologous SCT and then undergo allogeneic SCT on day 0. Patients receive GM-CSF as in autologous SCT.
* Post-SCT imatinib mesylate therapy: After recovery from autologous or allogeneic SCT, patients receive oral imatinib mesylate once daily. Imatinib mesylate therapy continues in the absence of disease progression or unacceptable toxicity.

  * Group II (Ph chromosome-negative patients):
* Intensification therapy: Beginning 4 weeks after the completion of the second induction therapy, patients receive high-dose MTX IV over 2 hours on days 1, 8, and 22; leucovorin calcium IV every 6 hours for 4 doses and then orally every 6 hours for 12 doses beginning 22-24 hours after each MTX infusion; and ASP IV over 30 minutes on days 2, 9, and 23.

Patients who are ≤ 50 years of age with a histocompatible donor proceed to allogeneic SCT and undergo allogeneic SCT as in group I. Patients who are ≤ 50 years of age without an appropriate donor are randomized to 1 of 2 treatment arms.

* Arm I (conventional consolidation/maintenance therapy):

  * Conventional consolidation therapy: During course 1, patients receive ARA-C IV over 30 minutes and VP-16 IV over 1 hour on days 1-5; VCR IV on days 1, 8, 15, and 22; and oral dexamethasone on days 1-28. During course 2 (which begins 4 weeks after initiation of course 1 or when blood counts recover), patients receive ARA-C and VP-16 as in course 1. During course 3 (which begins 4 weeks after initiation of course 2 or when blood counts recover), patients receive DNR IV on days 1, 8, 15, and 22; CTX IV over 30 minutes on day 29; ARA-C IV over 30 minutes on days 31-34 and 38-41; and oral thioguanine on days 29-42. During course 4 (which begins 8 weeks after initiation of course 3 or when blood counts recover), patients receive treatment as in course 2.
  * Maintenance therapy: Beginning 4 weeks after initiation of course 4 of consolidation therapy or when blood counts recover, patients receive oral MP daily; MTX orally or IV once weekly; VCR IV once every 12 weeks; and oral PRED for 5 days every 12 weeks. Maintenance therapy continues for 2.5 years after initiation of intensification therapy.
* Arm II (autologous SCT): Patients undergo autologous SCT as in group I with the exception of high-dose consolidation/mobilization chemotherapy.

Patients are followed every 6 months for 2 years.

PROJECTED ACCRUAL: Approximately 40 patients per year will be accrued for group I (Philadelphia [Ph] chromosome-positive patients) of this study. Approximately 550 patients will be accrued for group II (Ph chromosome-negative patients) of this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute lymphoblastic leukemia (ALL)

  * More than 25% lymphoblasts in bone marrow

    * Patients with myeloid antigen expression AND unequivocal lymphoid immunophenotype are eligible
* Philadelphia (Ph) chromosome status determined by cytogenetics, fluorescence in situ hybridization (FISH), and/or RNA analysis

  * Patients determined to be Ph chromosome negative by cytogenetics, but positive for BCR-ABL by FISH or polymerase chain reaction are considered Ph chromosome positive
  * Patients with Ph chromosome-positive disease may be up to age 65
* No myelodysplasia or other antecedent hematologic disorder
* Patients age 50 and under must be HLA typed during induction therapy of study treatment OR provide a written explanation for not undergoing HLA typing

  * A and B typing required
  * C and DR typing done if feasible
* Allogeneic stem cell transplantation patients must meet the following criteria:

  * Appropriate HLA histocompatible donor available

    * Ph chromosome-negative patients must have HLA identical sibling
    * Ph chromosome-positive patients must have HLA identical, HLA-matched unrelated, or haploidentical related donor
* Postinduction therapy:

  * CSF negative for leukemia
  * No occult or overt leukemic meningitis
  * Documented complete remission

PATIENT CHARACTERISTICS:

Age:

* 15 to 65

Performance status:

* Induction therapy:

  * Not specified
* Postinduction therapy:

  * 0-1

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Induction therapy:

  * Direct bilirubin ≤ 2.0 mg/dL
* Postinduction therapy:

  * Direct bilirubin < 2.0 mg/dL
  * SGPT or SGOT < 3 times normal

Renal:

* Induction therapy:

  * Creatinine < 2 mg/dL
* Postinduction therapy:

  * Creatinine ≤ 2 mg/dL
  * Creatinine clearance ≥ 60 mL/min

Cardiovascular:

* Induction and postinduction therapy:

  * No significant cardiac disease requiring digoxin and/or diuretics
  * No major ventricular dysrhythmia requiring medication
  * No ischemic heart disease requiring medication
* Postinduction therapy:

  * Cardiac ejection fraction ≥ 50% for patients under consideration for transplantation

Pulmonary:

* Induction therapy:

  * Not specified
* Postinduction therapy:

  * FEV_1 ≥ 60% of predicted for patients under consideration for transplantation
  * DLCO ≥ 50% of predicted for patients under consideration for transplantation

Other:

* Induction and postinduction therapy:

  * HIV negative
  * No concurrent organ damage or other medical problem (e.g., psychiatric disorder or drug abuse) that would preclude study therapy
  * Not pregnant
* Postinduction therapy:

  * No persistent infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent umbilical cord allogeneic transplantation

Chemotherapy:

* Not specified

Endocrine therapy:

* Prior corticosteroids for ALL allowed

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Induction and postinduction therapy:

  * No other prior therapy for ALL
* Postinduction therapy:

  * No concurrent antibiotics

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1929 (Actual)
Dates: Start 1993-05-07 (Actual); Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival | All patients were followed for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jacob M. Rowe, MD, Study Chair — Rambam Health Care Campus; Mark R. Litzow, MD, Principal Investigator — Mayo Clinic; Antony H. Goldstone, FRCP, Study Chair — University College London Hospitals
Locations (94):
- United States (94):
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Jewish Hospital Cancer Center, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College of Medicine - Center City Hahnemann Campus, Philadelphia, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin

REFERENCES:
- [Background] Wang H, Chen XQ, Geng QR, Liu PP, Lin GN, Xia ZJ, Lu Y. Induction therapy using the MRC UKALLXII/ECOG E2993 protocol in Chinese adults with acute lymphoblastic leukemia. Int J Hematol. 2011 Aug;94(2):163-168. doi: 10.1007/s12185-011-0891-y. Epub 2011 Jul 6. PMID 21732037
- [Background] Goldstone AH. Transplants in Adult ALL--? Allo for everyone. Biol Blood Marrow Transplant. 2009 Jan;15(1 Suppl):7-10. doi: 10.1016/j.bbmt.2008.11.017. PMID 19147069
- [Background] Ramanujachar R, Richards S, Hann I, Goldstone A, Mitchell C, Vora A, Rowe J, Webb D. Adolescents with acute lymphoblastic leukaemia: outcome on UK national paediatric (ALL97) and adult (UKALLXII/E2993) trials. Pediatr Blood Cancer. 2007 Mar;48(3):254-61. doi: 10.1002/pbc.20749. PMID 16421910
- [Background] Paietta E, Ferrando AA, Neuberg D, Bennett JM, Racevskis J, Lazarus H, Dewald G, Rowe JM, Wiernik PH, Tallman MS, Look AT. Activating FLT3 mutations in CD117/KIT(+) T-cell acute lymphoblastic leukemias. Blood. 2004 Jul 15;104(2):558-60. doi: 10.1182/blood-2004-01-0168. Epub 2004 Mar 25. PMID 15044257
- [Background] Ferrando AA, Neuberg D, Dodge RK, et al.: Adult T-cell ALL patients whose lymphoblasts express the HOX11 oncogene have an excellent prognosis when treated with chemotherapy and are not candidates for allogeneic bone marrow transplantaton in first remission. [Abstract] Blood 100 (11 pt 1): A-578, 2002.
- [Result] Moorman AV, Schwab C, Ensor HM, Russell LJ, Morrison H, Jones L, Masic D, Patel B, Rowe JM, Tallman M, Goldstone AH, Fielding AK, Harrison CJ. IGH@ translocations, CRLF2 deregulation, and microdeletions in adolescents and adults with acute lymphoblastic leukemia. J Clin Oncol. 2012 Sep 1;30(25):3100-8. doi: 10.1200/JCO.2011.40.3907. Epub 2012 Jul 30. PMID 22851563
- [Result] Sive JI, Buck G, Fielding A, Lazarus HM, Litzow MR, Luger S, Marks DI, McMillan A, Moorman AV, Richards SM, Rowe JM, Tallman MS, Goldstone AH. Outcomes in older adults with acute lymphoblastic leukaemia (ALL): results from the international MRC UKALL XII/ECOG2993 trial. Br J Haematol. 2012 May;157(4):463-71. doi: 10.1111/j.1365-2141.2012.09095.x. Epub 2012 Mar 13. PMID 22409379
- [Result] Patel B, Rai L, Buck G, Richards SM, Mortuza Y, Mitchell W, Gerrard G, Moorman AV, Duke V, Hoffbrand AV, Fielding AK, Goldstone AH, Foroni L. Minimal residual disease is a significant predictor of treatment failure in non T-lineage adult acute lymphoblastic leukaemia: final results of the international trial UKALL XII/ECOG2993. Br J Haematol. 2010 Jan;148(1):80-9. doi: 10.1111/j.1365-2141.2009.07941.x. Epub 2009 Oct 26. PMID 19863538
- [Result] Fielding AK, Rowe JM, Richards SM, Buck G, Moorman AV, Durrant IJ, Marks DI, McMillan AK, Litzow MR, Lazarus HM, Foroni L, Dewald G, Franklin IM, Luger SM, Paietta E, Wiernik PH, Tallman MS, Goldstone AH. Prospective outcome data on 267 unselected adult patients with Philadelphia chromosome-positive acute lymphoblastic leukemia confirms superiority of allogeneic transplantation over chemotherapy in the pre-imatinib era: results from the International ALL Trial MRC UKALLXII/ECOG2993. Blood. 2009 May 7;113(19):4489-96. doi: 10.1182/blood-2009-01-199380. Epub 2009 Feb 24. PMID 19244158
- [Result] Mansour MR, Sulis ML, Duke V, Foroni L, Jenkinson S, Koo K, Allen CG, Gale RE, Buck G, Richards S, Paietta E, Rowe JM, Tallman MS, Goldstone AH, Ferrando AA, Linch DC. Prognostic implications of NOTCH1 and FBXW7 mutations in adults with T-cell acute lymphoblastic leukemia treated on the MRC UKALLXII/ECOG E2993 protocol. J Clin Oncol. 2009 Sep 10;27(26):4352-6. doi: 10.1200/JCO.2009.22.0996. Epub 2009 Jul 27. PMID 19635999
- [Result] Marks DI, Paietta EM, Moorman AV, Richards SM, Buck G, DeWald G, Ferrando A, Fielding AK, Goldstone AH, Ketterling RP, Litzow MR, Luger SM, McMillan AK, Mansour MR, Rowe JM, Tallman MS, Lazarus HM. T-cell acute lymphoblastic leukemia in adults: clinical features, immunophenotype, cytogenetics, and outcome from the large randomized prospective trial (UKALL XII/ECOG 2993). Blood. 2009 Dec 10;114(25):5136-45. doi: 10.1182/blood-2009-08-231217. PMID 19828704
- [Result] Goldstone AH, Richards SM, Lazarus HM, Tallman MS, Buck G, Fielding AK, Burnett AK, Chopra R, Wiernik PH, Foroni L, Paietta E, Litzow MR, Marks DI, Durrant J, McMillan A, Franklin IM, Luger S, Ciobanu N, Rowe JM. In adults with standard-risk acute lymphoblastic leukemia, the greatest benefit is achieved from a matched sibling allogeneic transplantation in first complete remission, and an autologous transplantation is less effective than conventional consolidation/maintenance chemotherapy in all patients: final results of the International ALL Trial (MRC UKALL XII/ECOG E2993). Blood. 2008 Feb 15;111(4):1827-33. doi: 10.1182/blood-2007-10-116582. Epub 2007 Nov 29. PMID 18048644
- [Result] Paietta E, Li X, Richards S, et al.: Implications for the use of monoclonal antibodies in future adult ALL trials: analysis of antigen expression in 505 B-lineage (B-Lin) ALL patients (pts) on the MRC UKALLXII/ECOG2993 Intergroup trial. [Abstract] Blood 112 (11): A-1907, 2008.
- [Result] Patel B, Richards SM, Rowe JM, Goldstone AH, Fielding AK. High incidence of avascular necrosis in adolescents with acute lymphoblastic leukaemia: a UKALL XII analysis. Leukemia. 2008 Feb;22(2):308-12. doi: 10.1038/sj.leu.2405032. Epub 2007 Nov 8. PMID 17989709
- [Result] Rowe JM, Buck G, Moorman AV, et al.: Standard consolidation/maintenance chemotherapy is consistently superior to a single autologous transplant for adult patients with acute lymphoblastic leukemia: results of the international ALL trial (MRC UKALL XII/ECOG E2993). [Abstract] Blood 112 (11): A-3314, 2008.
- [Result] Fielding AK, Richards SM, Chopra R, Lazarus HM, Litzow MR, Buck G, Durrant IJ, Luger SM, Marks DI, Franklin IM, McMillan AK, Tallman MS, Rowe JM, Goldstone AH; Medical Research Council of the United Kingdom Adult ALL Working Party; Eastern Cooperative Oncology Group. Outcome of 609 adults after relapse of acute lymphoblastic leukemia (ALL); an MRC UKALL12/ECOG 2993 study. Blood. 2007 Feb 1;109(3):944-50. doi: 10.1182/blood-2006-05-018192. Epub 2006 Oct 10. PMID 17032921
- [Result] Fielding AK, Richards SM, Lazarus HM, et al.: Does imatinib change the outcome in Philapdelphia chromosome positive acute lymphoblastic leukaemia in adults? Data from the UKALLXII/ECOG2993 study. [Abstract] Blood 110 (11): A-8, 2007.
- [Result] Juric D, Lacayo NJ, Ramsey MC, Racevskis J, Wiernik PH, Rowe JM, Goldstone AH, O'Dwyer PJ, Paietta E, Sikic BI. Differential gene expression patterns and interaction networks in BCR-ABL-positive and -negative adult acute lymphoblastic leukemias. J Clin Oncol. 2007 Apr 10;25(11):1341-9. doi: 10.1200/JCO.2006.09.3534. Epub 2007 Feb 20. PMID 17312329
- [Result] Moorman AV, Harrison CJ, Buck GA, Richards SM, Secker-Walker LM, Martineau M, Vance GH, Cherry AM, Higgins RR, Fielding AK, Foroni L, Paietta E, Tallman MS, Litzow MR, Wiernik PH, Rowe JM, Goldstone AH, Dewald GW; Adult Leukaemia Working Party, Medical Research Council/National Cancer Research Institute. Karyotype is an independent prognostic factor in adult acute lymphoblastic leukemia (ALL): analysis of cytogenetic data from patients treated on the Medical Research Council (MRC) UKALLXII/Eastern Cooperative Oncology Group (ECOG) 2993 trial. Blood. 2007 Apr 15;109(8):3189-97. doi: 10.1182/blood-2006-10-051912. Epub 2006 Dec 14. PMID 17170120
- [Result] Lazarus HM, Richards SM, Chopra R, Litzow MR, Burnett AK, Wiernik PH, Franklin IM, Tallman MS, Cook L, Buck G, Durrant IJ, Rowe JM, Goldstone AH; Medical Research Council (MRC)/National Cancer Research Institute (NCRI) Adult Leukaemia Working Party of the United Kingdom and the Eastern Cooperative Oncology Group. Central nervous system involvement in adult acute lymphoblastic leukemia at diagnosis: results from the international ALL trial MRC UKALL XII/ECOG E2993. Blood. 2006 Jul 15;108(2):465-72. doi: 10.1182/blood-2005-11-4666. Epub 2006 Mar 23. PMID 16556888
- [Result] Rowe JM, Buck G, Burnett AK, Chopra R, Wiernik PH, Richards SM, Lazarus HM, Franklin IM, Litzow MR, Ciobanu N, Prentice HG, Durrant J, Tallman MS, Goldstone AH; ECOG; MRC/NCRI Adult Leukemia Working Party. Induction therapy for adults with acute lymphoblastic leukemia: results of more than 1500 patients from the international ALL trial: MRC UKALL XII/ECOG E2993. Blood. 2005 Dec 1;106(12):3760-7. doi: 10.1182/blood-2005-04-1623. Epub 2005 Aug 16. PMID 16105981
- [Result] Goldstone AH, Lazarus HJ, Richards SM, et al.: The outcome of 551 1st CR transplants in adult ALL from the UKALL XII/ECOG 2993 study. [Abstract] Blood 104 (11): A-615, 2004.
- [Result] Lazarus HM, Richards SM, Chopra R, et al.: Adult patients with acute lymphoblastic leukemia (ALL) and central nervous system (CNS) leukemia at diagnosis may attain durable complete remissions (CR). Results from the International ALL Trial (MRC UKALL-XII/ECOG E2993) . [Abstract] Blood 104 (11): A-4484, 2004.
- [Result] Goldstone AH, Chopra R, Buck G, et al.: The outcome of 267 Philadelphia positive adults in the international UKALL12/ECOG E 2993 study. Final analysis and the role of allogeneic transplant in those under 50 years. [Abstract] Blood 102 (11 Pt 1): A-268, 2003.
- [Result] Ferrando AA, Neuberg D, Dodge RK, et al.: Adult T-cell ALL patients whose lymphoblasts express the HOX11 oncogene have an excellent prognosis when treated with chemotherapy and are not candidates for allogeneic bone marrow transplantaton in first remission. [Abstract] Blood 100 (11 pt 1): A-578, 2002.
- [Result] Paietta E, Kim H, Racevskis J, et al.: Immunophenotypic characteristics, but not age or secondary cytogenetic changes, affect response and survival of BCR/ABL positive adult acute lymphoblastic leukemia (ALL): ECOG/MRC Intergroup trial, E2993. [Abstract] Blood 100 (11 pt 1): A-2990, 2002.
- [Result] Goldstone AH, Prentice HG, Durrant J, et al.: Allogeneic transplant (related or unrelated donor) Is the preferred treatment for adult Philadelphia chromosome positive (Ph+) acute lymphoblastic leukaemia (ALL). Results from the international ALL trial (MRC UKALLXII/ECOG E2993). [Abstract] Blood 98 (11 Pt 1): A-3556, 2001.
- [Result] Paietta E, Kim H, Rowe JM, et al.: Prognostic significance of immunophenotyping and cytogenetics in adult acute lymphoblastic leukemia (ALL): interim analysis of ECOG/MRC phase III intergroup trial, E2993. [Abstract] Blood 98 (11 Pt 1): A-3494, 2001.
- [Result] Rowe JM, Richards SM, Burnett AK, et al.: Favorable results of allogeneic bone marrow transplantation (BMT) for adults with Philadelphia (Ph)-chromosome-negative acute lymphoblastic leukemia (ALL) in first complete remission (CR): results from the international ALL trial (MRC UKALL XII/ECOG E2993). [Abstract] Blood 98 (11 Pt 1): A-2009, 2001.
- [Result] Goldstone AH, Richards S, Wiernik PH, et al.: Philadelphia chromosome positive patients with adult acute lymphoblastic leukemia (ALL). Early results from the international ALL trial. [Abstract] Blood 94 (suppl 1): 3071a, 1999.
- [Result] Rowe JM, Richards S, Wiernik PH, et al.: Allogenic bone marrow transplantation (BMT) for adults with acute lymphoblastic leukemia (ALL) in first complete remission (CR): early results from the international ALL trial. [Abstract] Blood 94 (suppl 1): 732a, 1999.
- [Result] Paietta E, Racevskis J, Neuberg D, Rowe JM, Goldstone AH, Wiernik PH. Expression of CD25 (interleukin-2 receptor alpha chain) in adult acute lymphoblastic leukemia predicts for the presence of BCR/ABL fusion transcripts: results of a preliminary laboratory analysis of ECOG/MRC Intergroup Study E2993. Eastern Cooperative Oncology Group/Medical Research Council. Leukemia. 1997 Nov;11(11):1887-90. doi: 10.1038/sj.leu.2400836. PMID 9369422
- [Derived] Fielding AK, Rowe JM, Buck G, Foroni L, Gerrard G, Litzow MR, Lazarus H, Luger SM, Marks DI, McMillan AK, Moorman AV, Patel B, Paietta E, Tallman MS, Goldstone AH. UKALLXII/ECOG2993: addition of imatinib to a standard treatment regimen enhances long-term outcomes in Philadelphia positive acute lymphoblastic leukemia. Blood. 2014 Feb 6;123(6):843-50. doi: 10.1182/blood-2013-09-529008. Epub 2013 Nov 25. PMID 24277073
- [Derived] Van Vlierberghe P, Ambesi-Impiombato A, De Keersmaecker K, Hadler M, Paietta E, Tallman MS, Rowe JM, Forne C, Rue M, Ferrando AA. Prognostic relevance of integrated genetic profiling in adult T-cell acute lymphoblastic leukemia. Blood. 2013 Jul 4;122(1):74-82. doi: 10.1182/blood-2013-03-491092. Epub 2013 May 17. PMID 23687089
- [Derived] Marks DI, Moorman AV, Chilton L, Paietta E, Enshaie A, DeWald G, Harrison CJ, Fielding AK, Foroni L, Goldstone AH, Litzow MR, Luger SM, McMillan AK, Racevskis J, Rowe JM, Tallman MS, Wiernik P, Lazarus HM. The clinical characteristics, therapy and outcome of 85 adults with acute lymphoblastic leukemia and t(4;11)(q21;q23)/MLL-AFF1 prospectively treated in the UKALLXII/ECOG2993 trial. Haematologica. 2013 Jun;98(6):945-52. doi: 10.3324/haematol.2012.081877. Epub 2013 Jan 24. PMID 23349309